CLINICAL TRIAL: NCT05910814
Title: The Effect of an Acute Bout of Physical Exercise on the Consolidation Phase of Motor Learning Acquired Through Physical or Mental Practice
Brief Title: Effect of Physical Exercise on Motor Learning Acquired With Physical or Mental Practice
Acronym: EPICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL22_0425; 2023-A00155-40 (Other: ID-RCB)
Record Dates: First submitted 2023-05-30; First posted 2023-06-20 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Physical Exercise; Motor Learning
Keywords: motor imagery; consolidation; BDNF; sleep deprivation; physical exercise
MeSH Terms: conditions — Motor Activity; Sleep Deprivation | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 6 arms will be enrolled, with 12 participants per group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PP (physical practice) (Experimental): Acquired the motor sequence physically
  Interventions: Behavioral: Normal Night (Night); Behavioral: Rest control; Behavioral: Physical Practice (PP)
- MI (motor imagery) (Experimental): Acquired the motor sequence mentally during training
  Interventions: Behavioral: Normal Night (Night); Behavioral: Rest control; Behavioral: Motor imagery
- MI+HIIE (motor imagery + high-intensity interval physical exercise) (Experimental): Acquired the motor sequence mentally and achieve a HIIE before the consolidation
  Interventions: Behavioral: Normal Night (Night); Behavioral: Physical Exercise (HIIE); Behavioral: Motor imagery
- PP+HIIE (physical practice + motor imagery + high-intensity interval physical exercise) (Experimental): Acquired the motor sequence physically and achieve a HIIE before the consolidation
  Interventions: Behavioral: Normal Night (Night); Behavioral: Physical Exercise (HIIE); Behavioral: Physical Practice (PP)
- SD + PP (sleep deprivation + physical practice) (Experimental): One night of sleep deprivation prior physical motor acquisition with PP and consolidation
  Interventions: Behavioral: Sleep Deprivation (SD); Behavioral: Rest control; Behavioral: Physical Practice (PP)
- SD+PP+HIIE (sleep deprivation + physical practice + high-intensity interval physical exercise) (Experimental): One night of sleep deprivation prior physical motor acquisition and HIIE before consolidation
  Interventions: Behavioral: Sleep Deprivation (SD); Behavioral: Physical Exercise (HIIE); Behavioral: Physical Practice (PP)

INTERVENTIONS:
Behavioral: Sleep Deprivation (SD) — Participants in the sleep deprivation group will spend a night awake, under the supervision of an investigator, at Croix-Rousse Hospital. The investigator will provide a list of activities to maintain the participant awake.
  Arms: SD + PP (sleep deprivation + physical practice); SD+PP+HIIE (sleep deprivation + physical practice + high-intensity interval physical exercise)
Behavioral: Normal Night (Night) — Participants in the normal night group will spend one night sleeping in their own home.
  Arms: MI (motor imagery); MI+HIIE (motor imagery + high-intensity interval physical exercise); PP (physical practice); PP+HIIE (physical practice + motor imagery + high-intensity interval physical exercise)
Behavioral: Physical Exercise (HIIE) — Participants in the physical exercise group (i.e. IM+HIIE, PP+HIIE, SD+PP+HIIE) will start with a 2-minute warm-up on an ergometer cycle.
  After the warm-up, they will perform 3 minutes of exercise at a workload customized to their maximal aerobic power (MAP) corresponding to 80 % their MAP and then rest actively for 2 minutes at 40 % of MAP. This cycle of 5 minutes will be repeated 3 times in row, resulting in a total of 17 minutes of physical exercise including the warm-up.
  Arms: MI+HIIE (motor imagery + high-intensity interval physical exercise); PP+HIIE (physical practice + motor imagery + high-intensity interval physical exercise); SD+PP+HIIE (sleep deprivation + physical practice + high-intensity interval physical exercise)
Behavioral: Rest control — Participants will watch a documentary during an equivalent time as the physical exercise (i.e. 17 minutes).
  Arms: MI (motor imagery); PP (physical practice); SD + PP (sleep deprivation + physical practice)
Behavioral: Motor imagery — On the bimanual finger tapping task composed of 8 elements, the participant will be required to repeat the motor sequence mentally using MI (mental rehearsal of movement) during twelve blocks of 30 seconds. Participant will imagine performing the sequence as fast and accurately as possible without overt movement.
  Arms: MI (motor imagery); MI+HIIE (motor imagery + high-intensity interval physical exercise)
Behavioral: Physical Practice (PP) — Participants will practice a bimanual sequential finger tapping task composed of 8 movements. Participant will be required to perform the sequence as fast and as accurately as possible during blocs of 30 s (i.e. twelve blocs during training).
  Arms: PP (physical practice); PP+HIIE (physical practice + motor imagery + high-intensity interval physical exercise); SD + PP (sleep deprivation + physical practice); SD+PP+HIIE (sleep deprivation + physical practice + high-intensity interval physical exercise)

SUMMARY:
Motor learning is crucial for human daily routine, involving the acquisition of new movements. It consists of an online acquisition phase followed by offline consolidation, where motor memory is organized into stable representations. Acquisition can be achieved through physical practice (PP, overt repetition of movement) or mental rehearsal using motor imagery (MI). Recent studies suggest that high-intensity interval physical exercise (HIIE) enhances motor learning, particularly during consolidation, by promoting neural plasticity mediated by brain-derived neurotrophic factor (BDNF). However, the impact of HIIE on sequential motor consolidation with PP or MI remains poorly understood.

In contrast, sleep deprivation (SD) reduces BDNF release and neural plasticity. Limited research has explored the effects of SD on motor acquisition, especially sequential motor learning. Considering the opposing effects of HIIE and SD, performing HIIE after SD may protect motor consolidation processes.

This study aims to examine the influence of HIIE on sequential motor learning using PP or MI under both sleep-deprived and normal sleep conditions. Six groups, each comprising 12 participants, will learn an 8-item bimanual sequence.

* MI group: acquired the motor sequence mentally during training
* MI+HIIE group: acquired the motor sequence mentally and achieve a HIIE before the consolidation
* PP: acquired the motor sequence physically
* PP+HIIE group: acquired the motor sequence physically and achieve a HIIE before the consolidation
* SD+PP group: one night of sleep deprivation prior physical motor acquisition with PP and consolidation
* SD+PP+HIIE group: one night of sleep deprivation prior physical motor acquisition and HIIE before consolidation.

All groups will be tested on the sequence at the beginning and the end of the acquisition phase (pre- and post-acquisition), and after the physical exercise (i.e. HIIE) or the rest period (post-exercise).

Hypothesis of this study are :

* Acute physical exercise (HIIE) would enhance the consolidation of motor memory (post-exercise) after physical and mental acquisition (PP,MI) compared to conditions without exercise.
* One night of sleep deprivation would affect the acquisition and consolidation of motor learning.

Physical exercise would compensate for the detrimental effects of sleep deprivation on the consolidation of motor learning.

DETAILED DESCRIPTION:
The ability to learn new movement (i.e. motor learning) is an essential part of the human daily routine. Motor learning is typically characterized by an online acquisition phase followed by an offline consolidation phase (i.e., without further practice) whereby the motor memory traces are reorganized into stable and long-lasting representations. The acquisition can be achieved through physical practice (PP, overt repetition of the movement) or through motor imagery (MI, covert rehearsal of movement). Over the last two decades, studies have demonstrated that performing high intensity interval exercise (HIIE) can enhance motor learning and particularly the consolidation phase. It seems that HIIE induced a favourable physiological cascade that contributes to the neural plasticity. In this vein, both lactate and brain derived neurotrophic factor (BDNF) biological markers seems to play a major role in long-term memory consolidation. To date, little is known on the HIIE contribution to sequential motor consolidation with PP or MI.

By contrast to HIIE, sleep deprivation decreased the BDNF released and the neural plasticity. There are very few studies that have examined the impact of sleep deprivation (SD) on motor acquisition and only one on sequence motor learning. Considering the antagonistic effects of HIIE and SD, it might possible that performing HIIE following SD could protect the motor consolidation processes.

Therefore, the main goal of this study is to understand the influence of HIIE on sequential motor learning through PP or MI under condition of sleep deprivation and normal night. In this study, six groups will be enrolled each including 12 participants. All groups will learn a bimanual sequence of 8 items.

* MI group: acquired the motor sequence mentally during training
* MI+HIIE group: acquired the motor sequence mentally and achieve a HIIE before the consolidation
* PP: acquired the motor sequence physically
* PP+HIIE group: acquired the motor sequence physically and achieve a HIIE before the consolidation
* SD+PP group: one night of sleep deprivation prior physical motor acquisition with PP and consolidation
* SD+PP+HIIE group: one night of sleep deprivation prior physical motor acquisition and HIIE before consolidation.

All groups will be tested on the sequence at the beginning and the end of the acquisition phase (pre- and post-acquisition), and after the physical exercise (i.e. HIIE) or the rest period (post-exercise).

Hypothesis of this study are :

* Acute physical exercise (HIIE) would enhance the consolidation of motor memory (post-exercise) after physical and mental acquisition (PP,MI) compared to conditions without exercise.
* One night of sleep deprivation would affect the acquisition and consolidation of motor learning.
* Physical exercise would compensate for the detrimental effects of sleep deprivation on the consolidation of motor learning.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 35
* Available for the entire study (13 days maximum)
* Right-handed upper limbs with a score > 0.5 on the Edinburgh laterality test
* Having dated and signed an informed consent
* Subject affiliated or entitled to a social security scheme
* Absence of contraindication to the practice of physical activity
* Considered active according to the GPAQ (Global Physical Activity Questionnaire)
* Neutral or moderate circadian typology (31 to 69)
* Regular physical activity (2h/week minimum)

Exclusion Criteria:

* Musculoskeletal injury < 6 months
* Pathology or surgical intervention resulting in a locomotor disorder < 6 months
* Chronic or disabling neurological, cardiovascular or psychic pathology
* Resting heart rate > 100 bpm
* Pittsburgh Sleep Quality Index > 10
* Taking sleeping pills or medication with a psychoactive effect during the last 6 months
* Ongoing participation in an interventional research
* Pregnant or breastfeeding women
* Person deprived of judicial or administrative freedom.
* Contraindication to TMS (Transcranial Magnetic Stimulation):
* Frequent or severe headaches
* History of epilepsy
* Head trauma with loss of consciousness
* Implanted equipment (including implanted pacemaker or defibrillator, cochlear implant, pump administering medication, surgical clips, metal shrapnel)
* Neurosurgical intervention (in particular eye surgery)
* An open wound on the scalp
* Consumption of more than three glasses of alcohol per day

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Number of correct sequence between post-acquisition and post-exercise for PP and PP+HIIE | Through study completion, an average of 13 days.
  In the bimanual finger tapping task, the accuracy corresponds to the number correct sequence performed during a block of practice The primary outcome measure will be the difference in the number of correct sequences performed between the end of acquisition (post-acquisition) and consolidation (post-exercise) stages between the PP and PP+HIIE.

SECONDARY OUTCOMES:
Number of correct sequence between post-acquisition and post-exercise for IM and IM+HIIE | Through study completion, an average of 13 days.
  In the bimanual finger tapping task, the accuracy corresponds to the number correct sequence performed during a block of practice.
  This secondary outcome measure will be the difference in the number of correct sequences performed between the end of acquisition (post-acquisition) and consolidation (post-exercise) stages between the IM and IM+HIIE.
Number of correct sequence between pre-acquisition, post-acquisition, and post-exercise for SD and SD+PP | Through study completion, an average of 13 days.
  In the bimanual finger tapping task, the accuracy corresponds to the number correct sequence performed during a block of practice.
  This secondary outcome measure will be the difference in the number of correct sequences performed between the beginning of the acquisition (pre-acquisition), the end of acquisition (post-acquisition) and the consolidation (post-exercise) stages between the SD and SD+PP groups.
Number of correct sequence between post-acquisition and post-exercise for SD+PP and SD+PP+HIIE | Through study completion, an average of 13 days.
  In the bimanual finger tapping task, the accuracy corresponds to the number correct sequence performed during a block of practice.
  This secondary outcome measure will be the difference in the number of correct sequences performed between the end of acquisition (post-acquisition) and consolidation (post-exercise) stages between the SD+PP and SD+PP+HIIE groups.
Neurophysiological informations between pre-acquisition, post-acquisition and post-exercise for all groups (IM, PP, IM+HIIE, PP+HIIE, SD+PP, SD+PP+HIIE) | Through study completion, an average of 13 days.
  Neurophysiological measurement will be collected with transcranial magnetic stimulation (TMS). TMS is a tool that generate a magnetic field that depolarizes the neuron in primary motor cortex and offers the opportunity to probe the cortico-spinal excitability (CSE) through motor evoked potential (MEP).
  To consider the muscle fibers excitability when analysing MEP amplitude, responses will be normalized to the maximal M-wave. The assessment of M-wave for the first dorsal interosseous muscle will be achieved with a single constant-current stimulation applied on the ulnar nerves via a 30-mm anode-cathode bipolar felt pad.
  The average of MEP will be normalised to M wave using this formula :
  MEP normalised=((Mean MEP (mV))/(Mean Mmax (mV) ))*100 The MEP Normalised will be compared for all groups between the three-time frame pre-acquisition, post-acquisition and post-exercise
BDNF assessment between pre-acquisition and post-exercise for all groups | Through study completion, an average of 13 days.
  Biological variables will include the measurement of three molecules: lactate, BDNF and cortisol.
  A 5 ml blood sample will be collected from an antecubital vein and will be immediately centrifuged. The plasma will be separated from the serum and stored at -80 °C. BDNF(brain-derived neurotrophic factor) levels will be analysed by means of enzyme-linked immunosorbent assay method (ELISA Kit) at the end of study.
  BDNF will be compared for all groups between the two-time frames pre-acquisition and post-exercise
Lactate assessment between pre-acquisition and post-exercise for all groups | Through study completion, an average of 12 days.
  Biological variables will include the measurement of three molecules: lactate, BDNF and cortisol.
  Blood lactate will be collected from a capillary blood on the finger and will be immediately analysed using a lactate analyser device.
  Lactate will be compared for all groups between the two-time frames pre-acquisition and post-exercise
Cortisol assessment between pre-acquisition and post-exercise for all groups | Through study completion, an average of 13 days.
  Biological variables will include the measurement of three molecules: lactate, BDNF and cortisol.
  A 5 ml blood sample will be collected from an antecubital vein and will be immediately centrifuged. The plasma will be separated from the serum and stored at -80 °C. Cortisol levels will be analysed by means of enzyme-linked immunosorbent assay method (ELISA Kit) at the end of study.
  Cortisol will be compared for all groups between the two-time frames pre-acquisition and post-exercise
Number of correct sequence between post-acquisition and post-exercise for PP and MI groups | Through study completion, an average of 13 days.
  In the bimanual finger tapping task, the accuracy corresponds to the number correct sequence performed during a block of practice.
  This secondary outcome measure will be the difference in the number of correct sequences performed between the end of acquisition (post-acquisition) and consolidation (post-exercise) stages between the PP and MI groups.
Number of correct sequence between post-acquisition and post-24h for all groups | Through study completion, an average of 13 days.
  In the bimanual finger tapping task, the accuracy corresponds to the number correct sequence performed during a block of practice.
  This secondary outcome measure will be the difference in the number of correct sequences performed between the end of acquisition (post-acquisition) and the next day after a night's sleep (post-24h) for all groups.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime PINGON, MD, Principal Investigator — EFR-Médecine du sport et de l'activité physique, HCL
Locations (2):
- France (2):
  - Service d'explorations fonctionnelles respiratoires-Médecine du sport et de l'activité physique, Hôpital de la Croix-Rousse, Hospices Civils de Lyon, Lyon
  - Laboratoire LIBM, Université Lyon 1, Villeurbanne